CLINICAL TRIAL: NCT04717505
Title: Evaluation of Dual Task Performance in Rheumatic Diseases: A Case-Control Study
Brief Title: Dual Task Performance in Rheumatic Diseases
Status: Completed | Type: Observational
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Emel Taşvuran Horata, PhD; Assistant Professor, Afyonkarahisar Health Sciences University
Other Study IDs: 2020/513
Record Dates: First submitted 2021-01-14; First posted 2021-01-22 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Rheumatic Diseases
MeSH Terms: conditions — Rheumatic Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Control Group: Demographic information ( age, gender, occupation, weight, height) of all participants in the study will be recorded first. The cognitive functions of all participants within the scope of the study will be evaluated in the Standardized Mini Mental Test; The 10 Meter Walk Test for dual task assessments will be applied in 3 different ways, with a portable gait device with wearable sensors: 1-single task conditions, 2-dual task conditions (motor + cognitive), 3-dual task conditions (motor + motor).
  Interventions: Other: Gait Assessments; Other: Standardized Mini Mental Test
- Rheumatological Condition Group: Demographic information (diagnosis, age, gender, occupation, weight, height) of all participants in the study will be recorded first. The cognitive functions of all participants within the scope of the study will be evaluated in the Standardized Mini Mental Test; The 10 Meter Walk Test for dual task assessments will be applied in 3 different ways, with a portable gait device with wearable sensors: 1-single task conditions, 2-dual task conditions (motor + cognitive), 3-dual task conditions (motor + motor). In addition, in order to evaluate their health status, only the case group will be applied Arthritis Impact Measurement Scales 2 (questionnaire) and Visual Analogue Scale for pain assessment.
  Interventions: Other: Gait Assessments; Other: Arthritis Impact Measurement Scales 2; Other: Visual Analogue Scale; Other: Standardized Mini Mental Test

INTERVENTIONS:
Other: Gait Assessments — 10 Meter Walking Test: It is applied by walking at a normal walking speed (like walking in a shopping mall) without any assistance at a marked distance of 10 meters.
  1- Evaluation of walking under single task conditions is done with the 10 Meter Walk Test and without any cognitive or motor second task. Evaluation of walking under dual task conditions is applied in two different ways: 2-adding a cognitive task to the walking motor task (motor + cognitive dual task) 3-adding one more motor task to the walking motor task (motor + motor dual task). While performing dual tasks, the time-distance (walking speed, cadence, stride length) characteristics of the gait are recorded using with wearable gait device.
  Other Names: 10 meter Walking Test
Other: Arthritis Impact Measurement Scales 2 — It is a multidimensional, disease-specific, self-administered questionnaire designed to measure health status outcomes in patients with arthritis.
  Groups: Rheumatological Condition Group
Other: Visual Analogue Scale — The Visual Analogue Scale is a reliable and easily applicable scale used to measure the pain intensity of patients, accepted in the world literature.
  Groups: Rheumatological Condition Group
Other: Standardized Mini Mental Test — Although the test has limited specificity in terms of differentiating clinical syndromes, it is a short, useful and standardized method that can be used to determine the cognitive level globally.

SUMMARY:
Chronic pain is pain that exceeds the duration of the injury or trigger stimulus and lasts for at least three months. Recent studies show that chronic pain has devastating effects on cognitive functions by causing emotional stress, anxiety, and depression.The studies show that chronic pain affects certain cognitive areas. These areas are; processing speed, short-term memory, longterm memory, inhibitory control and working memory. In addition, task-oriented studies show that chronic pain affects not single tasks, but rather dual tasks that require the use of complex cognitive function (executive function). 40-60% of rheumatologic patients do not have sufficient relief in their pain. For this reason, dual task performance may be affected in individuals diagnosed with rheumatological disease, secondary to the impairment of cognition. In the literature, there are only limited studies showing dual-task performance effects in individuals diagnosed with fibromyalgia and osteoarthritis. However, chronic pain is the main health problem that prevents mobility restriction and participation in all rheumatic diseases. In addition, there is no study investigating the dual task performance effect in rheumatic diseases in a comprehensive way. Therefore, the aim of the study is to investigate the effect of rheumatic diseases on dual-task performance by comparing it with the control group.

DETAILED DESCRIPTION:
Pain is an unpleasant sensory or emotional experience associated with actual or potential tissue damage and is classified as acute or chronic. Acute pain is felt for a short time after an injury or harmful stimulus and is considered part of a defense strategy; It points to an active danger to the organism. Chronic pain that exceeds the duration of the injury or trigger stimulus and lasts for at least three months. Recent studies show that chronic pain has devastating effects on cognitive functions by causing emotional stress, anxiety, and depression. Studies show that chronic pain affects certain cognitive areas. These areas are; processing speed, short-term memory, long-term memory, inhibitory control and working memory. In addition, task-oriented studies show that chronic pain affects not simple tasks, but rather dual tasks that require the use of complex cognitive function (executive function).

Task; it is a behavior, skill or ability that needs to be done. The simple (single) task contains only one alert or task. For example, walking. Dual task requires the simultaneous performance of two different tasks that can be measured independently and have different goals. For example, calculating while walking at the same time. In rehabilitation approaches, single or dual task trainings are applied. Among physiotherapy and rehabilitation approaches, single task training consists only of exercises involving motor performance; Dual task trainings can consist of different exercise combinations that require two different tasks to be performed at the same time as motor + motor, cognitive + cognitive or motor + cognitive performances. The clinical benefit of dual task training is that most of the daily living activities are done in dual task conditions.

Chronic pain is a common health problem associated with most rheumatic diseases. It is pain that lasts for at least 3 months and cannot be completely relieved with standard pain medication. 40-60% of rheumatologic patients do not have sufficient relief in their pain. For this reason, dual-task performance may be affected in individuals diagnosed with rheumatological disease, secondary to the impairment of cognition. In the literature, there are only limited studies showing dual-task performance effects in individuals diagnosed with fibromyalgia and osteoarthritis. However, chronic pain is the main health problem that prevents mobility restriction and participation in all rheumatic diseases. In addition, there is no study investigating the dual task performance effect in rheumatic diseases in a comprehensive way. Therefore, the aim of thestudy is to investigate the effect of rheumatic diseases on dual-task performance by comparing it with the control group.

ELIGIBILITY:
Inclusion Criteria:

* For the case group

  * Having been diagnosed with any rheumatic disease (rheumatoid arthritis, ankylosing spondylitis… etc.) by a rheumatologist.
  * Not having any acute (fracture, surgery, etc.) or chronic disease (cognitive, neurological, etc.) other than rheumatic disease
  * Being in the age range of 18-65.
  * Presence of chronic pain for at least 3 months
  * Pain over 3.4 cm according to the Visual Analogue Scale (having moderate pain).
  * Standardized Mini Mental Test score> 24
  * At least primary education or literacy
* For control group:

  * Absence of any known acute (fracture, surgery, etc.) or chronic disease (cognitive, neurological, etc.)
  * Being in the age range of 18-65
  * Standardized Mini Mental Test score> 24
  * Having at least primary education or literacy

Exclusion Criteria:

* Both control and case groups

  * The presence of any problems (physical, cognitive or psychological) that will prevent the evaluations to be applied within the scope of the research
  * Being pregnant

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: For case group: Patients who come to Afyonkarahisar Health Sciences University Hospital Rheumatology Outpatient Clinic for treatment will constitute the case group of the study.
  For control group: Healthy individuals working in Afyonkarahisar Health Sciences University will constitute the control group of the study.
Sampling Method: Non-Probability Sample
Enrollment: 75 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Gait Speed | 10 minutes
  The time it takes to walk a specified distance
Cadence | 10 minutes
  Number of steps per minute
Step lengths | 10 minutes
  Step length is the distance between the point of initial contact of one foot and the point of initial contact of the opposite foot.

CONTACTS AND LOCATIONS:
Overall Officials: EMEL TAŞVURAN HORATA, Principal Investigator — Afyonkarahisar Health Science University
Locations (1):
- Afyonkarahisar Health Science University, Afyonkarahisar, Turkey (Türkiye)